CLINICAL TRIAL: NCT04841798
Title: Monoamine Oxidase B Occupancy in Depressed Patients
Brief Title: MAO-B Occupancy in Depressed Patients
Acronym: MOCP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: REB#094/2018
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Major Depressive Disorder; Treatment Resistant Depression
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Duloxetine (Other): Assessment of MAO-B distribution volume in the prefrontal cortex before and after duloxetine at 60 mg daily.
  Interventions: Other: [11C]SL25.1188 PET radiotracer
- Rasagiline (Other): Assessment of regional MAO-B distribution volume before and after rasagiline at 1.0 mg daily.
  Interventions: Other: [11C]SL25.1188 PET radiotracer
- Tranylcypromine (Other): Assessment of regional MAO-B distribution volume before and after tranylcypromine at 30 to 60 mg daily.
  Interventions: Other: [11C]SL25.1188 PET radiotracer

INTERVENTIONS:
Other: [11C]SL25.1188 PET radiotracer — Monoamine oxidase B (MAO-B) occupancy before and after medication treatment using [11C]SL25.1188 PET

SUMMARY:
The study is looking at assessing monoamine oxidase B (MAO-B) occupancy in depressed patients before and after medication treatment using positron emission tomography (PET) scan.

DETAILED DESCRIPTION:
BACKGROUND

1.1 Problem of Treatment Resistant Depression and a Proposed Solution

Problem of Major Depressive Disorder: Major depressive disorder (MDD) known to the layperson as clinical depression, is an illness composed of repeated major depressive episodes of variable length and persistence (MDE).

MDD is the leading cause of death and disability in moderate to high income countries. MDD is common with 5% of adults in the midst of a major depressive episode (MDE) and the lifetime prevalence of MDD is 10 to 20%. MDD is also often treatment resistant, with 50% of people having inadequate responses. Plausible Mechanism of Treatment Resistance: It is generally believed that there are multiple underlying pathologies in MDD and the mismatch of treatment to pathology results in treatment resistance. Hence it is important to determine whether common brain pathologies are targeted by common treatments like serotonin and norepinephrine reuptake inhibitors, and to establish the degree to which alternative treatments might better target such brain pathologies. Then with this information matching of treatment to identified disease pathologies can be optimized.

STUDY OBJECTIVES

Overview Rationale for Objectives The abnormal elevation in MAO-B level in MDE of MDD was most prominent in the prefrontal cortex, hence the investigators prioritize this region in our objectives. As detailed in the introduction, the investigators will assess MAO-B occupancy of tranylcypromine because it is a MAO-B inhibitor, albeit non-selective, that is approved in Canada for clinical use to treat MDD. The investigators assess rasagiline as a selective MAO-B inhibitor that does not require stringent dietary restriction of tyramine at the 1mg dose, which is approved for Parkinson's Disease in Canada and has potential to be purposed to treat MDD. The investigators will also include assessment of MAO-B VT before and after duloxetine to verify the widespread assumption that the commonly prescribed medications that inhibit the reuptake of serotonin and norepinephrine, do not affect MAO-B level.

Primary Objectives

1. To measure MAO-B occupancy of tranylcypromine at a standard treating dose (30 to 60mg total per day) in the prefrontal cortex.
2. To measure MAO-B occupancy of rasagiline at 1mg total daily, a dose not requiring stringent tyramine dietary restriction in the prefrontal cortex.

   Secondary Objective
3. To evaluate the effect of duloxetine 60mg daily on MAO-B VT in the prefrontal cortex.
4. To evaluate the relationship between changes in symptoms of MDE and cognition (primarily assessed with the Hamilton Rating Scale and the Cognitive Failure Questionnaire) and baseline MAO-B VT in the regions most altered in MDE, and MDE post COVID-19.

The methods to quantitate more exact occupancy inherently require some MAO-B occupancy to occur, so in the case of objective 3, the related measure of change in MAO-B VT will be assessed. In addition, investigators will evaluate MAO-B occupancy of the interventions listed in objectives 1 and 2 within other brain regions with either reasonably high MAO-B density or whose dysfunction is implicated in the pathophysiology of MDD, including the anterior cingulate cortex, ventral striatum, dorsal striatum, thalamus, hippocampus, and midbrain. With respect to objective 4, it is expected that participants with more elevated MAO-B VT will have a greater response to rasagiline.

ELIGIBILITY:
Inclusion Criteria:

* age 18 to 80
* DSM-5 diagnosis of current MDE and MDD verified by the research version of SCID for DSM-5
* early onset type MDD with first MDE prior to age 40
* score greater than or equal to 17 on the 17 item Hamilton Depression Rating Scale (HDRS)28
* antidepressant free for at least 2 weeks (by self report)
* worsening of MDE symptoms or new onset MDE symptoms after COVID-19 may receive rasagiline and complete all procedures except the second [11-C]SL25.1188 PET scan - participants with this criteria will be enrolled in the alternative criteria that is similar to the general criteria except for the second PET scan.

Exclusion Criteria:

* history of psychotic symptoms
* history of antisocial or borderline personality disorders (screened with the Structured Clinical Interview for Personality Disorders (SCID) for Diagnostic and Statistical Manual-5 (DSM-5) (unless occuring after COVID)
* history of neurodegenerative illness
* cigarette smoking for the past 6 months (there are reports that cigarette smoking lowers monoamine oxidase B 31, 32.)
* currently abusing street drugs
* current alcohol use disorder
* diagnosis of liver or kidney disease
* positive for hepatic dysfunction as measured by aspartate transaminase (AST) and alanine transaminase (ALT) tests
* diagnosis of cardiovascular disease such as hypertension/hypotension, angina or tachycardia
* electroconvulsive therapy or mechanical brain stimulation treatment within the previous 6 months (the effects of these on MAO-B level are unknown but since they could stimulate astrogliosis which could influence MAO-B level these are included as exclusionary)
* positive pregnancy test (in our Centre women up to 65 years of age are given a urine pregnancy test prior to every PET scan)
* currently breastfeeding
* recent use of MAO-B inhibitor treatments (within the previous 4 weeks)
* disorders of coagulation, blood or ongoing use of anticoagulant medication
* presence of metal objects or implanted electrical devices in the body that would preclude MRI scanning
* claustrophobia
* weight over 400lbs and height over 7ft (requirements for fitting in the scanners and hospital gowns)
* the total radiation dose over the currently approved guideline of 20 millisievert (mSv) in a 12-month period. Note: The sievert is a derived unit of ionizing radiation dose in the International System of Units (SI) and is a measure of the health effect of low levels of ionizing radiation on the human body.
* history of undergoing a number of PET scans that, including the number of PET scans under this protocol, will bring the total to more than 8 PET scans/lifetime, exceeding permissible limit for subjects participating in research set by our centre's guidelines
* elevated liver transaminases AST and ALT levels as shown by the laboratory test results

Additional Requirements for Receiving Tranylcypromine :

* not taking any anesthetics, meperidine (Demerol), anti-asthmatics, anti-hypertensives, dextromethorphan, buspirone, narcotics, codeine (e.g. found in Tylenol), over the counter medication for colds, hay fever, sinus decongestants, eye drops that contain tetrahydrozoline hydrochloride (Visine); SSRI medication including selective reuptake inhibitors (SSRI), amitriptyline, nortriptyline, protriptyline, desipramine, imipramine, doxepin, perphenazine, carbamazepine, cyclobenzaprine, amoxapine, maprotiline, trimipramine; stimulant medication such as: amphetamines, ephedrine, cocaine, methylphenidate, methyldopa, dopamine, levodopa, tryptophan as well as energy-enhancing and weight-reducing preparations for at least 2 weeks
* not taking fluoxetine for at least 6 weeks
* inadequate response to serotonin reuptake inhibitor medication
* inadequate response to medication that raises norepinephrine
* inadequate response to lithium addition to an antidepressant or patient does not want to take lithium due to side effects (such as intention tremor or hypothyroidism risk)
* inadequate response to a medication that raises both serotonin and norepinephrine
* inadequate response to wellbutrin or participant is not able to take wellbutrin due to a contraindication or side effect or participant does not wish to take wellbutrin
* inadequate response to wellbutrin added to a second antidepressant or participant is not able to take wellbutrin due to a contraindication or side effect or participant does not wish to take wellbutrin
* awareness and willingness to follow medication and substance use requirements required of taking tranylcypromine or rasagiline

Exclusion

* previous hypersensitivity to monoamine oxidase inhibitors
* previous history of hypersensitivity to tyramine
* self report of previous diagnosis of cerebrovascular or cardiovascular disorders
* self report history of recurrent or frequent headaches
* diagnosis of phaeochromocytoma and catecholamine-releasing paragangliomas
* systolic blood pressure not between 91 and 139 mmHg (inclusive)
* diastolic blood pressure not between 51 and 90 mmHg (inclusive)
* a decrease in systolic blood pressure of 20 mm Hg or diastolic blood pressure of 10 mm Hg within three minutes of standing when compared with BP from the sitting position
* use of triptans or tryptamines (e.g. sumatriptan or rizatriptan) in the past 2 weeks.

Additional Requirements for Taking Rasagiline

Inclusion

● Participant does not wish to take tranylcypromine due to concerns regarding side effects or the strict dietary restrictions of reduced tyramine intake required for taking tranylcypromine.

Additional Requirements for Taking Duloxetine:

Inclusion

* Participants must be antidepressant free for at least 4 weeks prior to scanning (most antidepressants affect monoamines as does duloxetine so a longer period of being medication free is required to be able to separate effect of duloxetine from previous medication).
* Participant must not have a history of non-response to duloxetine at a daily dose of 60mg daily or higher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-03 (Actual)

PRIMARY OUTCOMES:
MAO-B occupancy of tranylcypromine at standard treating dose | 3 years
  MAO-B Occupancy is an overall occupancy measure that is intended to be derived from Lassen Plot. The Lassen Plot will include MAO-B total distribution volume (VT) values before and after treatment in regions that optimize the plot. It is expected that these will include prefrontal cortex, anterior cingulate cortex, dorsal putamen, ventral striatum, hippocampus, and cerebellum. To quantify the regional monoamine oxidase B (MAO-B) occupancy we use a measure called the total distribution volume (VT) an index of MAO-B density. The percent change, termed occupancy can range from 0% to 100%.
MAO-B occupancy of rasagiline at standard treating dose | 3 years
  MAO-B Occupancy is an overall occupancy measure that is intended to be derived from Lassen Plot. The Lassen Plot will include MAO-B total distribution volume (VT) values before and after treatment in regions that optimize the plot. It is expected that these will include prefrontal cortex, anterior cingulate cortex, dorsal putamen, ventral striatum, hippocampus, and cerebellum. To quantify the regional monoamine oxidase B (MAO-B) occupancy we use a measure called the total distribution volume (VT) an index of MAO-B density. The percent change, termed occupancy can range from 0% to 100%.

SECONDARY OUTCOMES:
Rasagiline effect on MAO-B distribution volume (VT) in the prefrontal cortex | 3 years
  Rasagiline effect on MAO-B distribution volume (VT) in the prefrontal cortex. To quantify the regional monoamine oxidase B (MAO-B) occupancy we use a measure called the total distribution volume (VT) an index of MAO-B density. The percent change, termed occupancy can range from 0% to 100%.
Rasagiline effect on MAO-B distribution volume (VT) and cognition in MDE post COVID-19 | 3 years
  Rasagiline effect on the total Hamilton Depression Rating Scale (HDRS). The Hamilton Rating Scale for Depression (HRSD) scoring is based on the 17-item scale. Scores of 0-7 are considered as being normal, 8-13 higher than normal, 14-16 modestly clinical, 17-19 mild depression, 20-23 moderate depression and scores 24 or greater are considered severe depression. The maximum sore being 52. Higher scores represent worse outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey H Meyer, MD, PhD, Principal Investigator — CAMH
Locations (1):
- CAMH, Toronto, Ontario, Canada